CLINICAL TRIAL: NCT03016507
Title: Intraocular Pressure Variation by Pneumatic Tonometer Before and After Phacoemulsification
Acronym: IPOFACO
Status: Completed | Type: Observational
Sponsor: VER Excelência em Oftalmologia (Other)
Collaborators: Francisco Welington Rodrigues (Unknown)
Responsible Party: Principal Investigator, Rodrigo Egidio da Silva, Ophtalmologist, VER Excelência em Oftalmologia
Other Study IDs: VEREO 3
Record Dates: First submitted 2017-01-06; First posted 2017-01-10 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Intraocular Pressure; Cataracts Senile
Keywords: intraocular pressure; phacoemulsification; cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objective of this study is to evaluate the IOP variation before and 30 days after performing phacoemulsification through pneumatic tonometry, in addition to evaluating the factors possibly related to this variation.

DETAILED DESCRIPTION:
Cataracts represent the major cause of treatable blindness in developing countries. According to data , there are 45 million blind people in the world, of which 40% is due to cataract etiology. In Brazil, there are about 350,000 individuals blinded by cataracts.

One of the consequences observed after the cataract surgery is the variation of intraocular pressure (IOP). IOP is directly related to the volume of aqueous humor in the anterior chamber. Reports of oscillations after a cataract surgery range from +1.3 to -2.5 mmHg. The duration of this oscillation varies according to the literature studied. Some studies show that the oscillation seen in the first postoperative year was maintained for the 10-year period and was similar in patients of all ages. However, other authors have identified a non-permanent oscillation, which makes this topic controversial in ophthalmology.

There are a number of factors related to the degree of IOP reduction after a cataract surgery. Studies have shown that the preoperative IOP value, the depth of the anterior chamber, the volume of irrigation used during surgery and the age of the patients may interfere with the IOP variation in the postoperative period.

However, the gold standard tonometer for IOP measurement is Goldmann's. This measurement is closely related to important characteristics of the cornea, such as its thickness and curvature, and may underestimate or overestimate IOP values.

Another way to measure IOP is through a non-contact tonometer, blow or pneumatic. The blow tonometer has a pneumatic system that produces a jet of air, which leads to flattening of the cornea and on the surface of which a beam of parallel light rays is projected, in which only the reflected parallel and coaxial rays are picked up by the receiver of the device, obtaining a maximum peak of light reception when the cornea is flattened. Its main advantage is in its use in screening programs, the need for the use of eye drops and the lowest rates of contamination. The blow tonometer, as well as the flattening tonometer, is influenced by corneal factors, such as curvature and thickness, presenting the same parameters of under and overestimation of IOP.

The objective of this study is to evaluate the IOP variation before and 30 days after performing phacoemulsification through pneumatic tonometry, in addition to evaluating the factors possibly related to this variation.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* deep anterior chamber visualized by the slit lamp with open angle estimation using the Van Herick technique
* IOP lower than 21 mmHg
* without surgical intercurrences, submitted to phacoemulsification

Exclusion Criteria:

* younger than 18 years
* shallow anterior chamber visualized by slit lamp with estimation of narrow angle
* preoperative surgical complications
* IOP greater than 21 mmHg
* contact lens wearers
* eye surgeries and/or ocular diseases and/or systemic disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with cataract and with good systemic health
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-07; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Intraocular Pressure Variation by Pneumatic Tonometer Before and After Phacoemulsification | Six months

CONTACTS AND LOCATIONS:
Locations (1):
- Rodrigo Egidio da Silva, Goiânia, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poley BJ, Lindstrom RL, Samuelson TW, Schulze R Jr. Intraocular pressure reduction after phacoemulsification with intraocular lens implantation in glaucomatous and nonglaucomatous eyes: evaluation of a causal relationship between the natural lens and open-angle glaucoma. J Cataract Refract Surg. 2009 Nov;35(11):1946-55. doi: 10.1016/j.jcrs.2009.05.061. PMID 19878828
- [Background] Poley BJ, Lindstrom RL, Samuelson TW. Long-term effects of phacoemulsification with intraocular lens implantation in normotensive and ocular hypertensive eyes. J Cataract Refract Surg. 2008 May;34(5):735-42. doi: 10.1016/j.jcrs.2007.12.045. PMID 18471626
- [Background] Slabaugh MA, Bojikian KD, Moore DB, Chen PP. The effect of phacoemulsification on intraocular pressure in medically controlled open-angle glaucoma patients. Am J Ophthalmol. 2014 Jan;157(1):26-31. doi: 10.1016/j.ajo.2013.08.023. Epub 2013 Oct 30. PMID 24182743
- [Background] Damji KF, Konstas AG, Liebmann JM, Hodge WG, Ziakas NG, Giannikakis S, Mintsioulis G, Merkur A, Pan Y, Ritch R. Intraocular pressure following phacoemulsification in patients with and without exfoliation syndrome: a 2 year prospective study. Br J Ophthalmol. 2006 Aug;90(8):1014-8. doi: 10.1136/bjo.2006.091447. Epub 2006 May 3. PMID 16672324
- [Background] Bigger JF, Becker B. Cataracts and primary open-angle glaucoma: the effect of uncomplicated cataract extraction on glaucoma control. Trans Am Acad Ophthalmol Otolaryngol. 1971 Mar-Apr;75(2):260-72. No abstract available. PMID 4933971
- [Background] Yang HS, Lee J, Choi S. Ocular biometric parameters associated with intraocular pressure reduction after cataract surgery in normal eyes. Am J Ophthalmol. 2013 Jul;156(1):89-94.e1. doi: 10.1016/j.ajo.2013.02.003. Epub 2013 Apr 28. PMID 23628350
- [Background] Vincent SJ, Vincent RA, Shields D, Lee GA. Comparison of intraocular pressure measurement between rebound, non-contact and Goldmann applanation tonometry in treated glaucoma patients. Clin Exp Ophthalmol. 2012 May-Jun;40(4):e163-70. doi: 10.1111/j.1442-9071.2011.02670.x. Epub 2011 Oct 20. PMID 21883774
- [Background] Shingleton BJ, Pasternack JJ, Hung JW, O'Donoghue MW. Three and five year changes in intraocular pressures after clear corneal phacoemulsification in open angle glaucoma patients, glaucoma suspects, and normal patients. J Glaucoma. 2006 Dec;15(6):494-8. doi: 10.1097/01.ijg.0000212294.31411.92. PMID 17106361